CLINICAL TRIAL: NCT04552054
Title: Preoperative Mixed Reality Technique Combined With Three-Dimensional Printing Navigational Template Guided Localizing Pulmonary Small Nodules : a Prospective, Unicenter, Randomized Study.
Brief Title: Mixed Reality Technique Combined With 3D Printing Navigational Template for Localizing Pulmonary Nodules
Acronym: MR&3D Local
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen-zhao ZHONG (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Wen-zhao ZHONG, Principal Investigator, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46783912
Record Dates: First submitted 2020-08-28; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-05

CONDITIONS: Video-assisted Thoracic Surgery; Lung Cancer; Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
Keywords: pulmonary nodule; localization; three-dimensional printing; mixed reality
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CT guided localization (Active Comparator): Computerized Tomography(CT)-guided percutaneous lung puncture staining marker localization
  Interventions: Device: Computerized Tomography guided localization
- MR+3D guided localization (Experimental): Mixed reality(MR)+3D printing-guided percutaneous lung puncture staining marker localization
  Interventions: Device: Mixed Reality+ 3D printing guided localization

INTERVENTIONS:
Device: Mixed Reality+ 3D printing guided localization — Researchers project a three-dimensional reconstructed image of the patient's chest through MR glasses, then overlay the virtual chest with the actual chest. Finally, researchers put the three-dimensional printing navigational template on the surface of the body to guide for percutaneous lung puncture localization.
  Arms: MR+3D guided localization
Device: Computerized Tomography guided localization — CT-guided percutaneous lung puncture staining marker localization.
  Arms: CT guided localization

SUMMARY:
This study evaluates the viability and accuracy of preoperative mixed reality technique combined with three-dimensional printing navigational template guided localizing pulmonary small nodules.

DETAILED DESCRIPTION:
Pulmonary wedge resection is one of the most common types of operations performed by thoracic surgeons, especially given that more and more patients with ground glass nodules are being detected recently. One of the most significant current discussion concerning wedge resection is nodule localization. At present, a commonly used localization method is the CT-guided percutaneous lung puncture methylene blue staining marker localization, but this method has two main disadvantages: 1. the methylene blue dye is easy to spread, affecting the intraoperative judgment of nodule position by surgeon; 2. patients often suffer additional CT radiation. Mixed reality (MR) technique aims to enhance the simple self-visual effect and facilitate visualization of the surrounding environment in any situation. The three-dimensional model can be visualized by MR technique through MR glasses. Investigators project a three-dimensional reconstructed image of the patient's chest through MR glasses, then overlay the virtual chest with the actual chest, and then use this as a guide for percutaneous lung puncture localization. At the same time, investigators design an three-dimensional printing navigational template based on the 3D reconstruction model and place it on the surface of the body to help to guide the localization. This study is designed to evaluates the viability and accuracy of preoperative mixed reality technique combined with 3D printing navigational template guided localizing pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* a maximum target lung nodule (one or more) diameter ≤20 mm
* a target nodule CTR <0·25 or a minimum distance from the outer edge of the nodule to the nearest pleural surface >10 mm if the target nodule CTR was >0·25.
* Plan to perform VATS lung wedge resection

Exclusion Criteria:

* Inability to comply with research protocols or research procedures
* Any unstable systemic disease (including active infections, uncontrolled high blood pressure, unstable angina, angina pectoris that has started within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] Level II ), cardiac infarction (6 months before enrollment), severe arrhythmia requiring medication, liver, kidney or metabolic disease
* Active bleeding; Inability to withstand lying flat; Inability to cooperate through breathing during puncture
* Pregnant or lactating women
* Other circumstances that the investigator believes are not suitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Puncture success rate of localization | During surgery
  The deviations of less than 2 cm between the lesion and the injected site was defined as successful localization.

SECONDARY OUTCOMES:
Time of localization | During surgery
  To evaluate the time of the localization in each groups. The investigators record the start and end time of localization respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No